CLINICAL TRIAL: NCT02440698
Title: Experiences With a Healthcare Professional-mediated Genetic Test for Personalized Nutrition
Brief Title: Experiences With a Genetic Test for Personalized Nutrition Test for Personalized Nutrition
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Toronto (Other)
Collaborators: Nutrigenomix Inc. (Industry)
Responsible Party: Principal Investigator, Ahmed El-Sohemy, Associate Professor, University of Toronto
Other Study IDs: 31523
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Genetic test for personalized nutrition

SUMMARY:
The investigators will use a web-based survey to collect data on individual attitudes and self-reported health behaviour changes following genetic testing for personalized nutrition. Participants (n=80) are employees of a large multi-national food company's R&D division located in Australia, Switzerland, USA and the UK. They underwent a genetic test for personalized nutrition in March 2015 that was offered at no cost through the company wellness program. A registered dietitian completed a pre-test consultation and disclosed the test results with DNA-based dietary advice. The test provided information on 7 components of diet and additional information on individual risk for gluten intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Completed a genetic test for personalized nutrition through company wellness program.

Exclusion Criteria:

* None.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants (n=80) are employees of a large multi-national food company's R&D division located in Australia, Switzerland, USA and the UK. They underwent a genetic test for personalized nutrition in March 2015 that was offered at no cost through the company wellness program.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Health behaviour change | 3 months
  Do individuals self-report beneficial changes to their diets or lifestyle as a result of the DNA-based dietary advice?

OTHER OUTCOMES:
Sharing of information | 3 months
  Do individuals share their genetic test results with another healthcare professional?
Recommendation | 3 months
  Would individuals recommend genetic testing for personalized nutrition through a healthcare professional to others?
Satisfaction | 3 months
  Do individuals report satisfaction with undergoing genetic testing for personalized nutrition?
Interest in future testing | 3 months
  Do individuals report a desire to receive DNA-based dietary advice for other components of diet that were not assessed in the genetic test they underwent?

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El-Sohemy, PhD, Principal Investigator — University of Toronto; Daiva Nielsen, PhD, Study Director — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada